# Statistical Analysis Plan



| Sponsor | Pfizer |
|---|---|
| Protocol Title: | An International, Prospective Registry Investigating the Natural History of Children with Achondroplasia |
| Protocol Number: | C4181001 |
| Premier Research PCN: | THEC17754 |
| Document Version: | Final, 1.0 |
| Document Date: | 12-June-2020 |

## **Approvals**

| Role | Signatures | Date (dd-Mmm-yyyy) |
|---|---|---|
| Biostatistician,<br>Premier Research | Print Name: PPD , PhD Sign Name: PPD DocuSigned by: PPD PPD | |
| Medical Director,<br>Pfizer | Print Name: PPD , MBBS, PhD Sign Name: PPD | 22-+VO-2020 |
| Biostatistician,<br>Pfizer | Print Name: PPD Sign Name: PPD | |





## **Document History**

Not applicable.



## **Table of Contents**

| App | provals | | 1 |
|---|---|---|---|
| Doo | cument | History | 2 |
| Tab | ole of C | Contents | 3 |
| List | t of Tal | oles | 4 |
| 1. | Ov | rerview | 5 |
| 2. | Stu | ndy Objectives and Endpoints | 5 |
| | 2.1. | Study Objectives | 5 |
| | 2.2. | Study Endpoints | 5 |
| | 2.2.1. | Safety Endpoints | 5 |
| | 2.2.2. | Efficacy Endpoints | 6 |
| | 2.2.3. | Anthropometric Endpoints | 6 |
| | 2.2.4. | Achondroplasia-Related Symptoms, Test, and Treatment | 9 |
| | 2.2.5. | Non-achondroplasia-Related Conditions of Medical Significance | 9 |
| 3. | Ov | rerall Study Design and Plan | 9 |
| | 3.1. | Overall Design | 10 |
| | CCI | | |
| | 3.3. | Study Population | 10 |
| | 3.4. | Treatments Administered | 10 |
| | 3.5. | Method of Assigning Subjects to Treatment Groups | 10 |
| | 3.6. | Blinding and Unblinding | 10 |
| | 3.7. | Schedule of Events | 10 |
| 4. | Sta | tistical Analysis and Reporting | 12 |
| | 4.1. | Introduction | 12 |
| | 4.2. | Data Snapshot and Data Monitoring | 12 |
| 5. | An | alysis Populations | 12 |
| 6. | Ge | neral Issues for Statistical Analysis | 13 |
| | 6.1. | Statistical Definitions and Algorithms | 13 |
| | 6.1.1. | Baseline | 13 |
| | 6.1.2. | Handling of Dropouts or Missing Data | 13 |
| | 6.1.3. | Analysis Visit Windows | 13 |
| | 6.1.4. | Pooling of Sites | 13 |
| | 6.1.5. | Derived Variables. | 13 |
| | 6.1.6. | Data Adjustments/Handling/Conventions | 14 |



| Sponsor Pfizer Protocol Number C4181001 | research/ |
|------------------------------------------------------|-------------|
| PCN Number THEC17754 6.1.7. COVID-19 | 14 |
| 7. Study Subjects and Demographics | |
| 7.1. Disposition of Subjects and Withdrawals | |
| 7.2. Protocol Violations and Deviations | |
| 7.3. Demographics and Other Baseline Characte | |
| 8. Analysis of the Anthropometric Endpoints | |
| 8.1. Height SDS | |
| 8.2. Difference between Arm Span and Standing | |
| 9. Safety Analysis | |
| 9.1. Related Symptoms, Tests, and Treatments | |
| 9.2. Non-Achondroplasia-Related Conditions of | |
| 9.3. Physical Examinations | _ |
| 9.4. Collection of Blood Sample and X-ray of k | nees17 |
| 9.5. Concomitant Medication | |
| 10. Changes from Planned Analysis | 17 |
| 11. Other Planned Analysis | 17 |
| 12. References | 18 |
| 13. Tables, Listings, and Figures | 18 |
| 13.1. Planned Table Descriptions | 18 |
| 13.2. Planned Listing Descriptions | 21 |
| 13.3. Planned Figure Descriptions | 23 |
| 14. Tables, Listings, and Listing Shells | 24 |
| 14.1. Standard Layout for all Tables, Listings, an | d Figures24 |
| Appendix 1: Premier Research Library of Abbreviation | ıs25 |
| Appendix 2: Calculation of the Height-for-Age SDS | 26 |
| List of Tables | |
| Table 1: Anthropometric Measurements | 6 |
| Table 2: Schedule of Events | 11 |
| Table 3: Demographic Data Summary Tables and Figu | res |
| Table 4: Anthropometric Data | |
| Table 5: Safety Data | |
| Table 6: Planned Listings | |
| Table 7: Planned Figures | 23 |

Statistical Analysis Plan,





#### 1. Overview

This master statistical analysis plan (SAP) describes the planned analysis and reporting for Pfizer protocol number C4181001 (An International, Prospective Registry Investigating the Natural History of Children with Achondroplasia), dated 31-Jan-2019, version 2.0.

This study uses a primary master SAP and may require supplemental SAPs as well. An advantage of this study design is its ability to answer questions that emerge during the course of the study<sup>1</sup>. Subsequent and supplemental SAPs - triggered by new research questions emerging after the initial master SAP - can be developed when enough data become available, including data from other studies, to analyze a particular research question not included in this master SAP.

Reference materials for this statistical plan include the protocol, the anthropometric manual, and the accompanying sample data collection documents. Operational aspects related to collection and timing of planned clinical assessments are not repeated in this SAP unless relevant to the planned analysis.

The structure and content of this SAP provide sufficient detail to meet the requirements identified by the Food and Drug Administration, European Medicines Agency, and International Conference on Harmonization of Technical Requirements for Registration of Pharmaceuticals for Human Use: Guidance on Statistical Principles in Clinical Trials<sup>2</sup>. All work planned and reported for this SAP will follow internationally accepted guidelines, published by the American Statistical Association<sup>3</sup> and the Royal Statistical Society<sup>4</sup>, for statistical practice.

The planned analyses identified in this SAP may be included in clinical study reports (CSRs), regulatory submissions, or future manuscripts.

The statistical plan described hereafter is an *a priori* plan. It will be submitted to file prior to any inferential or descriptive analysis of data pertaining to Pfizer's study C4181001.

## 2. Study Objectives and Endpoints

## 2.1. Study Objectives

To investigate the natural history of children with achondroplasia in terms of:

- anthropometric characteristics
- achondroplasia-related symptoms, tests, and treatments
- biomarkers of bone growth

## 2.2. Study Endpoints

## 2.2.1. Safety Endpoints

Not applicable.



## 2.2.2. Efficacy Endpoints

Not applicable.

## 2.2.3. Anthropometric Endpoints

## **2.2.3.1. Anthropometric Measurements**

Anthropometric measurements will be done at all study visits and measurement results will be reported in the electronic case report form (eCRF). Anthropometric measurements will be performed according to the study-specific Anthropometric Measurement Manual.

The anthropometric endpoints of the study include specific measurements assessed at every visit or yearly. Moreover, the anthropometric manual requires performing 3 valid measurements for all endpoints during a visit, with the exception of body weight.

**Table 1: Anthropometric Measurements** 

| Measurements | Unit | Age group | Visit | # of valid<br>measurements |
|---|---|---|---|---|
| Standing height | cm | ≥2 years | Every visit | 3 |
| Height in supine position | cm | <2 years | Every visit | 3 |
| Sitting height | cm | ≥2 years | Every visit | 3 |
| Crown-rump length | cm | <2 years | Every visit | 3 |
| Knee height | cm | All | Every visit | 3 |
| Head Circumference | cm | All | Every visit | 3 |
| Arm Span | cm | All | Every visit | 3 |
| Elbow extension angle | degrees | All | Every visit | 3 |
| Knee extension angle | degrees | All | Every visit | 3 |
| Body weight | kg | All | Every visit | 1 |
| Forehead Results | cm | All | Every visit | 3 |
| Top of nose results | cm | All | Every visit | 3 |
| Base of nose results | cm | All | Every visit | 3 |
| Waist circumference | cm | All | Yearly | 3 |
| Chest circumference | cm | All | Yearly | 3 |



## 2.2.3.2. Derived Anthropometric Endpoints

Five additional anthropometric endpoints will be derived:

•

## 1. Height Growth (HG)

$$HG_i = \frac{OH_i - OH_0}{RH_i - RH_0}$$

where:

OH<sub>i</sub> = Observed Height in cm at visit i

 $OH_0 = Observed Height in cm at baseline$ 

RH<sub>i</sub> = Achondroplasia Reference Height at i (Merker at al., 2018)<sup>9</sup>

 $RH_0$  = Achondroplasia Reference Height at baseline

HG will be calculated every 3 months after baseline.

## 2. Sitting height/standing height (%)

The ratio (%) between the sitting height and the standing height will be calculated for all subjects.

## 3. Arm span/standing height (%)

The ratio (%) between the arm span and the standing height will be calculated for all subjects.

## 4. Difference between arm span and standing height (cm)

The difference between the arm span and the standing height will be calculated as: arm span (cm) – standing height (cm)

## 5. Height Standard Deviation Score (SDS)

The SDS for a given height or length in cm will be calculated using the LMS method

$$SDS = \frac{\left(\frac{height in cm}{M}\right)^{L} - 1}{LS}, L \neq 0$$

$$SDS = \frac{1}{S} \ln \left( \frac{height in \, on}{M} \right), L = 0$$



where L, M, and S are the interpolated values between the neighbouring values from the standard tables corresponding to the gender and to the exact age of the child. If the month is missing in the date of birth then the SDS will be set to missing.

L, M, and S, provided in the standard tables, are the tabulated fitted values of Box-Cox power, median, and coefficient of variation corresponding to the standard population, respectively.

If L=1 the formula for calculating the SDS can be written as:

$$SDS = \frac{\text{observed value - median value of the reference population}}{\text{standard deviation value of the reference population}}$$

where the median value is M and the standard deviation is MxS.

The same method will be applied for both the standing height and the recumbent length.

## 4.1 SDS with reference to normal population

The height-for-age SDS with reference to the normal population will be calculated using the 'WHO Child Growth Standards' from birth to 5 years and the 'WHO Reference 2007 for boys and girls, 5-19 years' for children older than 5 years.

The tables of the WHO Child Growth Standards are accessible in electronic format at <a href="www.who.int/childgrowth/standards/en">www.who.int/childgrowth/standards/en</a>; and the tables of the WHO Reference 2007 can be found at <a href="www.who.int/growthref">www.who.int/growthref</a>.

The following datasets available from the WHO websites will be used:

- lhfa boys p exp.txt
- lhfa girls p exp.txt
- hfa boys perc WHO2007 exp.txt
- hfa\_girls\_perc\_WHO2007\_exp.txt

The WHO standard tables assume that L=1 for all ages.

All SDS for children below 24 months are length-based and height-based otherwise. This means for children aged below 24 months (<731 days) and measured standing, the height will be converted to recumbent length by adding 0.7 cm; and for children aged 24 months or above who are measured in recumbent position, the length will be converted to standing height by subtracting 0.7 cm.

4.2 SDS with reference to achondroplasia population



The height-for-age SDS with reference to the achondroplasia population will be calculated on tabulations of population means (M), standard deviations (MxS), and coefficient of variation (S) Merker at al. (2018)<sup>9</sup>. Descriptive statistics and fitted values of L, M, and S for age are summarized in Supporting Information Table 2<sup>9</sup>.

L, M, and S values for finer ages values (age in exact years) will be interpolated between the neighbouring table values. The Merker standard tables assume that L=1 for all ages.

The same method for the standing height and the recumbent length will be applied. No adjustment to convert standing height and recumbent length will be applied when calculating the SDS with reference to the achondroplasia population.

Appendix 2 shows the calculation of the SDS for 3 examples.

## 2.2.4. Achondroplasia-Related Symptoms, Test, and Treatment

Achondroplasia-related symptoms will be collected according to relevant body systems and severity (mild, moderate, and severe).

Achondroplasia-related tests and treatment are also collected in the eCRF.

After the initial report on an important medical symptom, test, or treatment, the investigator should follow-up on the severity status of the medical symptoms, determine whether the symptom is ongoing or is resolved, and assess the outcome of a potential treatment until the child's participation in the study has ended.

## 2.2.5. Non-achondroplasia-Related Conditions of Medical Significance

Information concerning the diagnosis of any non-achondroplasia-related conditions of medical significance, including start and stop dates, should be reported. Information may be provided by parent(s) / legal guardian(s) or by the child if this is applicable.

## 3. Overall Study Design and Plan

This is a registry study in children with achondroplasia, aged 0-10 years, to be conducted at multiple clinical centers in several countries. Childrens' information will be collected in the registry at baseline and at every 3-month interval visits, for a maximum of 5 years. There will be a Screening visit, a Baseline visit, 3-month interval visits, a yearly visit ( $\pm 3$  weeks), and a Final visit.

The children may continue study participation until:

- Growth plates are considered to have fused, defined as standing height gain less than 1 cm within the last 6 months
- The child has reached the end of puberty (Tanner Stage V)





- The child is enrolled in an interventional study
- The child has participated in the study for 5 years
- The child is considered lost to follow-up

## 3.1. Overall Design



The study will enroll participants in the following approximate proportions:

- 40% 0-5y
- 40% 5-10y
- 20% 10-15y

## 3.3. Study Population

Children between 0 years and 15 years of age with achondroplasia documented by clinical diagnosis.

## 3.4. Treatments Administered

No investigational treatment will be administered.

## 3.5. Method of Assigning Subjects to Treatment Groups

No investigational treatment will be administered.

## 3.6. Blinding and Unblinding

Not applicable.

#### 3.7. Schedule of Events

A detailed schedule of events for the study is provided in Table 2.



**Table 2: Schedule of Events** 

| | Screening Visit <sup>a</sup> | <b>Baseline Visit</b> | Every 3 Months <sup>c</sup> | Every year | Final Visit <sup>c,d</sup> |
|---|---|---|---|---|---|
| Procedure | (Visit 0) | (Visit 1)b | (±3 weeks) | (±3 weeks) | (±3 weeks) |
| Informed consent and assent (as applicable) | X | | | | |
| Eligibility criteria | X | X | | | |
| Demographics | X | | | | |
| Medical and surgical history | X | X | | | |
| Physical examination | | X | X | | X |
| Waist circumference | | X | | X | X |
| Genetic confirmation of achondroplasiae | | (X) | | | |
| Anthropometric measurements | | X | X | | X |
| Achondroplasia-related symptoms, tests, and interventions | | X | X | | X |
| Non-achondroplasia-related symptoms, tests, and treatments $^{\rm f}$ | | X | X | | X |
| Tanner stage of puberty <sup>g</sup> | | X | X | | X |
| Collection of blood sample <sup>h</sup> | | X | | X | X |

a. Within 1 month before Baseline visit.

b. Screening visit and Baseline visit can be combined, if applicable.

c. Visits are scheduled relative to the date of the Baseline visit.

d The Final visit is conducted after termination criteria are met or after a decision to withdraw the child from the study.

e. If not available in medical records, then the result of genetic testing should be available as soon as possible, but not later than at the Final Visit.

f. Any non-achondroplasia-related important medical conditions and any treatment based on the medical judgment of the investigator that may affect the child's growth trajectory.

g. Only for children  $\geq$ 7 years of age (providing the investigator confirms there is no suspicion of a diagnosis of precocious puberty).

h. Fasting blood sample for biomarker analyses is required to be drawn in the morning. Sampling can be done, e.g., at a separate visit in the clinic, in the home by a visiting nurse, or at a local laboratory, whatever is most convenient and appropriate for the child's well-being.





## 4. Statistical Analysis and Reporting

#### 4.1. Introduction

Data processing, tabulation of descriptive statistics, calculation of inferential statistics, and graphical representations will be performed primarily using SAS (release 9.4 or higher).

Continuous (quantitative) variable summaries will include the number of subjects (n) with non-missing values, number of missing values (if applicable), mean, standard deviation (SD), median, minimum, and maximum. Continuous variables may be classed into groups and analyzed as a categorical variable when appropriate.

Categorical (qualitative) variable summaries will include the number of subjects (n) with non-missing values, number of missing values, frequency, and percentage of subjects who are in the particular category or each possible value. In general, the denominator for the percentage calculation will be based upon the total number of subjects in the study population with non-missing data.

The minimum and maximum will be reported with the same degree of precision (i.e., the same number of decimal places) as the observed data. Measures of location (mean and median) will be reported to 1 degree of precision more than the observed data and measures of spread (SD) will be reported to 2 degrees of precision more than the observed data.

Percentages will be presented to 1 decimal place, unless otherwise specified.

## 4.2. Data Snapshot and Data Monitoring

Data snapshot will be performed on a regular basis. This SAP describes the analytical principles and statistical techniques to be employed for both data snapshots and final analysis.

The sponsor may also request additional analysis during the study to analyze a particular research question that emerges during the course of the study.

A data safety monitoring board will not be used in this study.

#### 5. Analysis Populations

All analyses will be conducted on all enrolled children. The enroll set includes consented, screened, and eligibility-verified children.

Data after procedures or treatments that may affect height growth will be excluded from the analysis of anthropometric parameters. The Sponsor will review the subject-level data on an ongoing basis, providing information about procedures or treatment that may affect growth velocity.





## 6. General Issues for Statistical Analysis

## 6.1. Statistical Definitions and Algorithms

#### 6.1.1. Baseline

The observation recorded at Baseline visit (Visit 1) will be used as the baseline observation for all calculations of change from baseline.

## 6.1.2. Handling of Dropouts or Missing Data

In general, no data will be imputed. Missing intermediate or final measurements of the anthropometric measurements will not be replaced by imputed values.

## 6.1.3. Analysis Visit Windows

As per the protocol, a window of  $\pm 3$  weeks is allowed for the follow-up visits (Visits 2 to 20), while the Screening visit is planned within 1 month before the Baseline visit.

Statistical analyses will be based on scheduled visits collected in the eCRF without further realignment.

## 6.1.4. Pooling of Sites

Sites will not be taken into account in the analyses. Therefore, the question of pooling of sites is not applicable.

#### 6.1.5. Derived Variables

The following derived and computed variables have been initially identified as important for the descriptive summaries:

- 1. Height Growth (HG)Height Standard Deviation Score (SDS) with reference to normal population
- 2. Height SDS with reference to achondroplasia population
- 3. Sitting height/standing height (%)
- 4. Arm span/standing height (%)
- 5. Difference between arm span (cm) and standing height (cm)
- 6. Change from baseline = (value at current timepoint value at baseline)
- 7. Average of valid anthropometric measurements. When it is required to perform 3 valid measurements, the average of the 3 will be used in descriptive summaries. If 1 or 2



valid measurement are missing, the average will include only non-missing values. If all 3 measurements are missing then the average will be missing as well.

#### 8. Age at baseline

Age at baseline = (date of informed consent - date of birth)/365.25

Age will be rounded using 2 decimal places. If the day of birth is missing, but the month and year are present, age will be calculated based on day 1 if the month and year match the month/year of informed consent, or 15 if not. If the month is missing, age will be set to missing.

## 9. Exact age at each visit

- $\circ$  Exact age in years = (date of visit date of birth)/365.25
- $\circ$  Exact age in month = (date of visit date of birth)/30.4375
- Exact age in days = (date of visit date of birth)

The exact age (2 decimal places if in months, 3 decimal places if in years) will be used to calculate the height-for-age SDS. The use of the 2 date variables (date of birth and date of visit) for calculating the exact age of the child is the recommended approach as best practice. If the day is missing for the date of birth, 15 will replace it, unless the month and year of birth match the month and year of informed consent in which case the first of the month will be used. If the month is missing for the date of birth, the exact age values and the height-for age SDS will be set to missing.

10. Age groups at each visit. Three age groups will be identified: <2 years, 2-10 years, and ≥10 years. Children may move from an age group to the next one during the study.

## 6.1.6. Data Adjustments/Handling/Conventions

All collected data will be presented in listings. Data not subject to analysis according to this plan will not appear in any tables or graphs but will be included only in the data listings.

#### 6.1.7. COVID-19

A Coronavirus Disease 2019 (COVID-19) Continuity Plan has been to mitigate the negative effects of the COVID-19 pandemic on the conduct of this natural history registry.

The impact of COVID-19 on this study and participants will be described in tables and listings, and in the CSR.

The following aspects will be summarized when due to COVID-19:

• Subject who early terminated the study





- Changes to visit windows to accommodate delays for some assessments
- Protocol deviations

The situation is rapidly evolving and further updates to the COVID-19 Continuity Plan and to this SAP are possible and likely.

## 7. Study Subjects and Demographics

## 7.1. Disposition of Subjects and Withdrawals

The total number of subjects for each one of the following categories will be presented in tables:

- Consented subjects
- Screened subjects and reason for screening failure
- Enrolled subjects
- Completed subjects and reason for completion
- Reasons for study discontinuation

In summary tables for disposition of subjects, a breakdown by gender will be given.

The reason given for screening failure will be summarized in a separate table for screen failures.

#### 7.2. Protocol Violations and Deviations

Protocol deviations will be listed.

## 7.3. Demographics and Other Baseline Characteristics

Summary statistics for exact age at the Baseline visit, gender, race, ethnicity, and achondroplasia familiarity will be presented by gender.

For the continuous variables, the number of non-missing values and the mean, SD, minimum, median, and maximum will be tabulated.

The number and percent of subjects reporting various medical and surgical histories, grouped by Medical Dictionary for Regulatory Activities (MedDRA) system organ class (SOC) and preferred term (PT) (coded using MedDRA v.20.0), will be tabulated by gender. Medical and surgical histories by SOC and PT will be sorted in order of descending frequency in the overall group of the SOC and then by descending frequency orders of the PT within each SOC.

#### 8. Analysis of the Anthropometric Endpoints

Descriptive summaries of the observed value and change from baseline will be calculated for the anthropometric endpoints. For continuous variables, number of non-missing values, number of





missing values, the mean, SD, minimum, median, and maximum will be tabulated by gender. Subgroup analysis will be performed by age group at each visit.

Angles are circular quantities and are usually described using polar coordinates since the arithmetic mean may not be appropriate. However, angles for elbow and knee extension measure the deviation from a completely straight elbow or knee and are not circular quantities. The elbow extension angle and the knee extension angle will be summarized using the same descriptive statistics described for other anthropometric endpoints.

Height growth, height SDS, ration between sitting and standing heights, and ratio between arm span and standing height will be plotted against age separately by gender.

#### 8.1. Height SDS

As a complementary descriptive analysis the height SDS will be analyzed using a Mixed Model for Repeated Measure (MMRM) based on the restricted maximum likelihood (REML) approach.

Although the SDS is calculated standardizing for age and gender, the model will include a fixed effect of gender (binary) and a random effect of age (continuous) and a random intercept for each subject.

An unstructured covariance structure will be used to model the within-subject errors. If the analysis fails to converge, simpler structures (e.g. spatial power, ante-dependent, first autoregressive) will be tested; the covariance structure converging to the best fit, as determined by Akaike's information criterion will be used. Only the final model will be included in the TLFs.

The main goal of this model is to characterize the within-subject variability, the between-subjects variability, and to address any residual effect of gender and age.

Moreover, predicted trajectories of height SDS over age will be presented in a plot separately by gender.

## 8.2. Difference between Arm Span and Standing Height

The difference between the arm span and the standing height will be analyzed using the methods described in Section 8.1.

## 9. Safety Analysis

## 9.1. Related Symptoms, Tests, and Treatments

The number and percent of subjects reporting symptoms related to achondroplasia will be tabulated by gender, body system, and severity. The number and percent of subjects for each test and treatment related to achondroplasia will be described by gender.





## 9.2. Non-Achondroplasia-Related Conditions of Medical Significance

The non-achondropasia-related conditions of medical significance will be listed.

## 9.3. Physical Examinations

The number and percent of subjects with normal, abnormal, and clinical significant results will be calculated for each body system by visit and gender.

## 9.4. Collection of Blood Sample and X-ray of knees

The number and percent of subjects with blood sample collection, X-Ray of knees, and tibiofemoral angles measured will be described by visit and gender. Descriptive summaries of the tibiofemoral angles will be calculated and presented in a table.

#### 9.5. Concomitant Medication

Concomitant medications will be summarized descriptively by anatomical therapeutical chemical (ATC) level 2 and PT and gender using counts and percentages.

Prior medications will be presented only in listings separately from concomitant medications. Medications that started prior to date of informed consent will be considered prior medications. Any medications continuing or starting post the date of informed consent will be considered concomitant. If a medication starts prior to the date of the informed consent and continues after the date of the informed consent, it will be considered both prior and concomitant.

Medications will be coded using ATC classification level 2 (WHO-DD v. March 2017).

## 10. Changes from Planned Analysis

No change have been planned.

## 11. Other Planned Analysis

Pubertal status for boys and girls will be described using number and percent of subjects reporting various categories by visit and age group at each visit. Only children ≥7 years of age will be included in the analysis, providing the investigator confirms there is no suspicion of a diagnosis of precocious puberty.

Descriptive summaries will be calculated for the biomarkers of bone growth. Longitudinal modeling of biomarkers of bone growth will done in a manner similar to modeling of anthropometric parameters. Additional analyses for the biomarkers of bone growth may be requested and described in a separate analysis plan.





## 12. References

- 1. Registries for Evaluating Patient Outcomes, 3rd edition. Informed Consent for Registries. In: Eds Gliklich RE, Dreyer NA, Leavy MB. Rockville (MD): Agency for Healthcare Research and Quality (US); 2014 Rockville (MD): Agency for Healthcare Research and Quality (US).
- 2. US Federal Register. (1998) International Conference on Harmonization; Guidance on Statistical Principles for Clinical Trials. Department of Health and Human Services: Food and Drug Administration [Docket No. 97D-0174]. Federal Register Volume 63, Number 179, pages 49583-49598. September 16, 1998.
- 3. ASA. (2016) Ethical Guidelines for Statistical Practice. Prepared by the Committee on Professional Ethics, April 2016. http://www.amstat.org/about/ethicalguidelines.cfm
- 4. RSS. (2014) The Royal Statistical Society: Code of Conduct, 2014. http://www.rss.org.uk/Images/PDF/join-us/RSS-Code-of-Conduct-2014.pdf.
- 5. de Onis M, Onyango AW, Van den Broeck J, Chumlea WC, Martorell R. Measurement and standardization protocols for anthropometry used in the construction of a new international growth reference. Food and Nutrition Bulletin 2004;25(Supplement 1):S27-36.
- 6. de Onis M, Garza C, Onyango AW, Martorell R, editors. WHO Child Growth Standards. Acta Paediatrica Supplement 2006;450:S5-S101.
- 7. WHO Child Growth Standards: length /height-for-age, weight-for-age, weight-for-length, weight-forheight and body mass index-for-age. Methods and development. Geneva, Switzerland: World Health Organization, 2006.
- 8. de Onis M, Onyango AW, Borghi E, Siyam A, Nishida C, Siekmann J. Development of a WHO growth reference for school-aged children and adolescents. Bulletin of the World Health Organization 2007;85:660-7.
- 9. Merker A, Neumeyer L, Hertel NT, Grigelioniene G, Mäkitie O, Mohnike K, Hagenäs L. Growth in achondroplasia: Development of height, weight, head circumference, and body mass index in a European cohort. Am J Med Genet A. 2018 Aug;176(8):1723-1734. doi: 10.1002/ajmg.a.38853. Epub 2018 Aug 2.

#### 13. Tables, Listings, and Figures

All listings, tables, and graphs will have a header showing the sponsor company name and protocol and a footer showing the version of SAS, the file name and path, and the source of the data (case report form [CRF] page or listing number).

#### 13.1. Planned Table Descriptions

The following are planned summary tables for protocol number C4181001. The table numbers and page numbers are placeholders only and will be determined when the tables are produced.





## **Table 3: Demographic Data Summary Tables and Figures**

| Table/Figure<br>Number | Population(s) | Table/Figure Title / Summary | Supporting<br>Listing |
|---|---|---|---|
| 14.1 Baseline a | 14.1 Baseline and Demographic Data Summary Tables | | |
| 14.1.1 | All Subjects | Subject Disposition | 16.2.1.1<br>16.2.1.2 |
| 14.1.2 | Screen Failures | Reason for Screen Failure | 16.2.1.3 |
| 14.1.3.1 | Enrolled Subjects | Summary of Demographics and Baseline Characteristics | 16.2.4.1 |
| 14.1.3.2 | Enrolled Subjects | Genetic Confirmation of Achondroplasia | 16.2.4.4 |
| 14.1.3.3 | Enrolled Subjects | Medical and Surgical History by System Organ Class and<br>Preferred Term | 16.2.4.2 |



## **Table 4: Anthropometric Data**

| Table Number | Population(s) | Table Title / Summary | Supporting<br>Listing |
|---|---|---|---|
| 14.2 Anthropometric Tables | | | |
| 14.2.1.1 | Enrolled Subjects | Standing Height in Children Aged ≥2 Years by Visit | 16.2.6.1 |
| 14.2.1.2 | Enrolled Subjects | Height in Supine Position in Children Aged <2 Years by Visit | 16.2.6.1 |
| 14.2.1.3 | Enrolled Subjects | Sitting Height in Children Aged ≥2 Years by Visit | 16.2.6.1 |
| 14.2.1.4 | Enrolled Subjects | Crow-rump Length in Children Aged <2 Years by Visit | 16.2.6.1 |
| 14.2.1.5 | Enrolled Subjects,<br>Age groups | Knee Height by Visit | 16.2.6.1 |
| 14.2.1.6 | Enrolled Subjects, Age groups | Head Circumference by Visit | 16.2.6.1 |
| 14.2.1.7 | Enrolled Subjects, Age groups | Arm Span by Visit | 16.2.6.1 |
| 14.2.1.8 | Enrolled Subjects,<br>Age groups | Elbow Extension Angle by Visit | 16.2.6.1 |
| 14.2.1.9 | Enrolled Subjects,<br>Age groups | Knee Extension Angle by Visit | 16.2.6.1 |
| 14.2.2 | Enrolled Subjects, Age groups | Body Weight by Visit | 16.2.6.2 |
| 14.2.3.1 | Enrolled Subjects,<br>Age groups | Cranial Series - Forehead Results by Visit | 16.2.6.3 |
| 14.2.3.2 | Enrolled Subjects, Age groups | Cranial Series - Top of Nose Results by Visit | 16.2.6.3 |
| 14.2.3.3 | Enrolled Subjects, Age groups | Cranial Series - Base of Nose Results by Visit | 16.2.6.3 |
| 14.2.4.1 | Enrolled Subjects,<br>Age groups | Waist Circumference by Visit | 16.2.6.4 |
| 14.2.4.2 | Enrolled Subjects, Age groups | Chest Circumference by Visit | 16.2.6.4 |
| 14.2.5.1.1 | Enrolled Subjects,<br>Age groups | Height Growth by Visit | 16.2.6.5 |
| 14.2.5.1.2 | Enrolled Subjects | Statistical Analysis of Height Growth: MMRM | 16.2.6.5 |
| 14.2.5.2 | Enrolled Subjects | Height Standard Deviation Score with Reference to Normal Population by Visit | 16.2.6.6 |
| 14.2.5.3 | Enrolled Subjects | Height Standard Deviation Score with Reference to<br>Achondroplasia Population by Visit | 16.2.6.6 |
| 14.2.5.4 | Enrolled Subjects,<br>Age groups | Ratio Between Sitting Height and Standing Height by Visit | 16.2.6.7 |
| 14.2.5.5 | Enrolled Subjects, Age groups | Ratio Between Arm Span and Standing Height by Visit | 16.2.6.7 |
| 14.2.6.1.1 | Enrolled Subjects, Age groups | Difference Between Arm Span and Standing Height Growth by Visit | 16.2.6.5 |
| 14.2.6.1.2 | Enrolled Subjects | Statistical Analysis of Height Growth: MMRM | 16.2.6.5 |



**Table 5: Safety Data** 

| Table Number | Population(s) | Table Title / Summary | Supporting<br>Listing |
|---|---|---|---|
| 14.3 Safety Da | ata | | |
| 14.3.6 Other S | Safety Data Sumn | nary Tables | |
| 14.3.6.1.1 | Enrolled Subjects | Achondroplasia-Related Symptoms by Body System and Severity | 16.2.7.1 |
| 14.3.6.1.2 | Enrolled Subjects | Achondroplasia-Related Tests | 16.2.7.2 |
| 14.3.6.1.3 | Enrolled Subjects | Achondroplasia-Related Treatments | 16.2.7.3 |
| 14.3.6.2 | Enrolled Subjects | Non-Achondroplasia-Related Conditions of Medical Significance | 16.2.7.4 |
| 14.3.6.3 | Enrolled Subjects | Abnormal and Clinically Significant Physical Examination<br>Results | 16.2.9.1 |
| 14.3.6.4.1 | Enrolled Subjects,<br>Age groups | Pubertal Status for Boys by Visit | 16.2.9.2 |
| 14.3.6.4.2 | Enrolled Subjects,<br>Age groups | Pubertal Status for Girls by Visit | 16.2.9.3 |
| 14.3.6.5 | Enrolled Subjects | Concomitant Medications by ATC Level 2 and Preferred Term | 16.2.9.4 |
| 14.3.6.6 | Enrolled Subjects | Blood Sample Collection and X-Ray of Knees | 16.2.9.5<br>16.2.9.6 |

## 13.2. Planned Listing Descriptions

The following are planned data and subject data listings for protocol number C4181001.

In general, 1 listing will be produced per CRF domain. All listings will be sorted by gender, site, and subject number. All calculated variables will be included in the listings.

In all listings a blank line will be placed between each subject. Within a data listing, if an item appears line after line (e.g., repetition of subject number), then only the first occurrence will be displayed.

In data listings, the information for a subject will be kept on 1 page if possible, rather than splitting a subject's information across pages.





## **Table 6: Planned Listings**

| Data Listing Number | Population | Data Listing Title / Summary |
|---|---|---|
| 16.2 Subject Data I<br>16.2.1 Subject Disc | Listings<br>ontinuation/Comple | tion |
| Listing 16.2.1.1 | All Subjects | Informed Consent and Assignment to Enrolled Population |
| Listing 16.2.1.2 | Enrolled Subjects | Study Completion Status |
| Listing 16.2.1.3 | Screen Failures | List of Reasons for Screening Failure |
| Listing 16.2.1.4 | All Subjects | Visit Dates |
| 16.2.2. Protocol De | viations | |
| Listing 16.2.2.1 | Enrolled Subjects | Major Protocol Deviations |
| 16.2.3 Exclusion from | om the Analysis of A | Anthropometric Parameters |
| Listing 16.2.3.1 | Enrolled Subjects | Exclusion from the Analysis of<br>Anthropometric Parameters |
| 16.2.4 Demographi | c and Other Baselin | ne Characteristics |
| Listing 16.2.4.1 | Enrolled Subjects | Demographic Data and Baseline<br>Characteristics |
| Listing 16.2.4.2 | Enrolled Subjects | Medical and Surgical History |
| Listing 16.2.4.3 | Enrolled Subjects | Prior Medications |
| Listing 16.2.4.4 | Enrolled Subjects | Genetic Confirmation of Achondroplasia |
| 16.2.6 Individual A | nthropometric Data | 1 |
| Listing 16.2.6.1 | Enrolled Subjects | Anthropometric Measurements |
| Listing 16.2.6.2 | Enrolled Subjects | Body Weight |
| Listing 16.2.6.3 | Enrolled Subjects | Anthropometric Measurements - Cranial Series |
| Listing 16.2.6.4 | Enrolled Subjects | Anthropometric Measurements of Waist and<br>Chest Circumference |
| Listing 16.2.6.5 | Enrolled Subjects | Annual Growth Velocity |
| Listing 16.2.6.6 | Enrolled Subjects | Height Standard Deviation Score |
| Listing 16.2.6.7 | Enrolled Subjects | Ratios: Sitting Height/Standing Height and<br>Arm Span/Standing Height |
| 16.2.7 Symptoms, T | Tests, and Treatmen | nts Listing |
| Listing 16.2.7.1 | Enrolled Subjects | Achondroplasia-Related Symptoms |
| Listing 16.2.7.2 | Enrolled Subjects | Achondroplasia-Related Tests |
| Listing 16.2.7.3 | Enrolled Subjects | Achondroplasia-Related Treatments |



| Data Listing Number | Population | Data Listing Title / Summary |
|---|---|---|
| Listing 16.2.7.4 | Enrolled Subjects | Non-Achondroplasia-Related Conditions for Clinical Relevance |
| 16.2.9 Other Clinica | l Observations and M | leasurements |
| Listing 16.2.9.1 | Enrolled Subjects | Physical Examination Results |
| Listing 16.2.9.2 | Enrolled Subjects | Pubertal Status for Boys |
| Listing 16.2.9.3 | Enrolled Subjects | Pubertal Status for Girls |
| Listing 16.2.9.4 | Enrolled Subjects | Concomitant Medications |
| Listing 16.2.9.5 | Enrolled Subjects | Blood Sample Collection |
| Listing 16.2.9.6 | Enrolled Subjects | BX-Ray of Knees |
| Listing 16.2.9.7 | Enrolled Subjects | List of Patients Who Were Affected by COVID-19 |

## 13.3. Planned Figure Descriptions

The following are planned summary figures for the study.

**Table 7: Planned Figures** 

| Figure Number | Population | Figure Title/Summary | Supporting listing |
|---|---|---|---|
| 14.2.1 | Enrolled | Height Growth by Age and Gender | 16.2.6.5 |
| 14.2.2 | Enrolled | Height Standard Deviation Scores by Age and Gender | 16.2.6.6 |
| 14.2.3 | Enrolled | Ratio between Sitting Height and Standing Height by Age t and Gender | 16.2.6.7 |
| 14.2.4 | Enrolled | Ratio between Arm Span and Standing Height by<br>Age and Gender | 16.2.6.7 |
| 14.2.5 | Enrolled | Predicted Height SDS by Age and Gender | |





## 14. Tables, Listings, and Listing Shells

## 14.1. Standard Layout for all Tables, Listings, and Figures

Table and listing shells are provided as a separate document.

Note that programming notes may be added if appropriate after each table, listing, and figure shell.

The final statistical tables will be produced in the format of the shells and will additionally include "double" page numbering in the format "page xx of yy." The first page numbering will count all pages of the document continuously and the second numbering will count the pages for each table separately. The final statistical output will be provided as fully bookmarked pdf file, including a table of contents.

No shells are provided for figures.





## **Appendix 1: Premier Research Library of Abbreviations**

| Abbreviation | Definition |
|--------------|----------------------------------------------|
| AGV | Annual Growth Velocity |
| ATC | anatomical therapeutic chemical |
| CRF | case report form |
| CSR | clinical study report |
| eCRF | electronic case report form |
| HG | height growth |
| MedDRA | Medical Dictionary for Regulatory Activities |
| N | Number |
| PT | preferred term |
| SAP | statistical analysis plan |
| SD | standard deviation |
| SDS | Standard Deviation Score |
| SOC | system organ class |
| WHO | World Health Organization |
| WHO-DD | World Health Organization Drug Dictionary |





## **Appendix 2: Calculation of the Height-for-Age SDS**

This section shows how to calculate the SDS for 3 subjects:

| Subject ID | 001 | 002 | 003 |
|---|---|---|---|
| Gender | Male | Male | Female |
| Date of birth | 15 Dec 2005 | 15 Dec 2015 | 15 Dec 2015 |
| Date of measurement | 04 Sep 2013 | 07 Jul 2017 | 25 Aug 2018 |
| Age in years | 7.721 | 1.561 | 2.694 |
| Age in months | 92.65 | 18.727 | 32.3285 |
| Age in days | 2820 | 570 | 984 |
| Height or Length in cm | 103.2 | 65.2 | 74.4 |
| Type of measure | Standing Height | Length in supine position | Length in supine position |

For Subject 003 aged <24 months, the length in supine position is converted to standing height by subtracting 0.7 cm. The standing height for Subject 003 is 73.7 cm. The estimated standing height will be used to calculate the SDS with reference to the WHO population, while the observed length in supine position will be used to estimate the SDS with reference to the Achondroplasia population.

The L, M, and S values corresponding to the neighbouring tables values are:

| | WHO Reference Population | | | | Merker Reference Population | | | |
|---|---|---|---|---|---|---|---|---|
| Subject ID | Age | L | M | S | Age | L | М | S |
| 001 | 92 months | 1 | 125.4545 | 0.04406 | 7.0 years | 1 | 95.8 | 0.039666 |
| | 93 months | 1 | 125.9104 | 0.04414 | 8.0 years | 1 | 99.6 | 0.041165 |
| 002 | 570 days* | 1 | 82.9759 | 0.0331 | 1.5 years | 1 | 69.8 | 0.032951 |
| | - | - | - | - | 2.0 years | 1 | 72.9 | 0.032922 |
| 003 | 984 days* | 1 | 92.433 | 0.03939 | 2.5 years | 1 | 74.3 | 0.37685 |
| | - | - | - | - | 3.0 years | 1 | 76.8 | 0.038220 |

<sup>\*</sup>For children aged 0-5 years, the WHO Standard Table provides age in days (0 to 1856) and there is no need for linear interpolation.





## The interpolated L, M, and S values and the SDSs are:

| | WHO Reference Population | | | | |
|---|---|---|---|---|---|
| Subject ID | Age | L | М | S | SDS |
| 001 | 92.65 months | 1 | 125.7503201 | 0.04411191 | -4.06525 |
| 002 | 570 days | 1 | 82.9759 | 0.0331 | -6.48984 |
| 003 | 984 days | 1 | 92.433 | 0.03939 | -5.14511 |
| | Merker Reference Population | | | | |
| Subject ID | Age | L | М | S | SDS |
| 001 | 7.721 years | 1 | 98.53880903 | 0.040746134 | 1.160922 |
| 002 | 1.561 years | 1 | 70.17556468 | 0.032947718 | -2.15194 |
| 003 | 2.694 years | 1 | 75.2702 | 0.038220 | -0.30250 |